CLINICAL TRIAL: NCT02047019
Title: A Multicenter, Randomized, Double-Blind, Monotherapy-Controlled Study of Nifedipine Gastrointestinal Therapeutic System and Candesartan Cilexetil in Combination Taken Orally for 8 Weeks in Adult Subjects With Essential Hypertension Who Are Inadequately Controlled on 16 mg Candesartan Cilexetil Monotherapy
Brief Title: Monotherapy-Controlled Study of Nifedipine Gastrointestinal Therapeutic System and Candesartan Cilexetil in Combination in Subjects With Essential Hypertension Inadequately Controlled on Candesartan Cilexetil
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: GPDC decided to terminate the study
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14727; 2012-004493-26 (EudraCT Number)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Drug combination; Nifedipine GITS; Candesartan Cilexetil; Hypertension; Combination therapy
MeSH Terms: conditions — Hypertension | interventions — candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Candesartan (Active Comparator): Treatment with 1 capsule and 2 tablets once daily in the morning for 8 weeks (Candesartan 16 mg, Placebo combination A, Placebo combination B)
  Interventions: Drug: Candesartan Cilexetil; Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) 30/16mg matching placebo; Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106)
- Nifedipine/Candesartan-30/16 (Experimental): Treatment with 1 capsule and 2 tablets once daily in the morning for 8 weeks (Candesartan placebo, Placebo combination A, Combination nifedipine / candesartan 30/16 mg)
  Interventions: Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106); Drug: Candesartan matching placebo
- Nifedipine/Candesartan-60/16 (Experimental): Treatment with 1 capsule and 2 tablets once daily in the morning for 8 weeks (Candesartan placebo, Placebo combination B, Combination nifedipine / candesartan 60/16 mg)
  Interventions: Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106); Drug: Candesartan matching placebo; Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) 30/16mg matching placebo

INTERVENTIONS:
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), 30/16 mg, tablet, orally, once daily
  Arms: Nifedipine/Candesartan-30/16
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), 60/16 mg, tablet, orally, once daily
  Arms: Nifedipine/Candesartan-60/16
Drug: Candesartan Cilexetil — Candesartan Cilexetil, 16 mg, capsule, orally, once daily
  Arms: Candesartan
Drug: Candesartan matching placebo — Candesartan matching placebo, capsule, orally, once daily
  Arms: Nifedipine/Candesartan-30/16; Nifedipine/Candesartan-60/16
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) 30/16mg matching placebo — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) 30/16mg matching placebo, tablet, orally, once daily
  Arms: Candesartan; Nifedipine/Candesartan-60/16
Drug: Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106) — Nifedipine GITS/Candesartan Cilexetil FDC(BAY98-7106), 60/16mg matching placebo, tablet, orally, once daily
  Arms: Candesartan; Nifedipine/Candesartan-30/16

SUMMARY:
This study examines the efficacy and safety of the Fixed Dose combination BAY98-7106 (nifedipine plus candesartan) in patients with hypertension, who do not achieve adequate control of blood pressure with candesartane alone.

Patients meeting the entry criteria, will receive candesartan alone 16mg in the first five weeks of the study to assess blood pressure control with candesartan given alone.

Patients with an insufficient therapeutic response to candesartan alone (defined by mean seated systolic blood pressure >/=140 mm/Hg) will enter the next part of the study, and will be randomly assigned to one of 3 treatments ( candesartan alone 16mg, combination nifedipine / candesartan 30/16 mg, combination nifedipine / candesartan 60/16 mg). Neither patient nor the treating physician will know which treatment is given (double-blinded design).This part of the study will last eight weeks.

ELIGIBILITY:
* Inclusion Criteria:
* Male and female subjects 18 years or older are eligible.
* At Visit 0, subjects not treated with antihypertensive medications are to have MSSBP (mean seated systolic blood pressure) of >/= 160 mmHg and < 200 mmHg, and 24 hours MASBP (mean ambulatory systolic blood pressure) >/= 130 mmHg; those subjects treated with antihypertensive medication are to have MSSBP >/= 150 mmHg and < 200 mmHg as measured by a calibrated electronic BP measuring device
* At Visit 3,subject must have MSSBP >/= 140 mmHg before randomization.
* Women of childbearing potential and men must agree to use adequate contraception other than hormonal contraceptives when sexually active. This applies since signing of the IC (informed consent)form until the last study drug administration.
* Exclusion Criteria:
* Mean seated systolic blood pressure (MSSBP) >/= 200 mmHg and/or mean seated diastolic blood pressure (MSDBP) >/= 120 mm/Hg
* Mean seated diastolic blood pressure (MSDBP) < 60 mm/Hg
* Differences greater than 20 mmHg for systolic blood pressure (SBP) and 10 mmHg for diastolic blood pressure (DBP) are present on 3 consecutive blood pressure readings at visit 0
* Evidence of secondary hypertension such as coarctation of the aorta, pheochromocytoma, hyperaldosteronism, etc.
* Cerebrovascular ischemic event (stroke, transient ischemic attack [TIA]) within the previous 12 months
* History of hypertensive retinopathy - known Keith-Wagener Grade III or IV. Any history of heart failure, New York Heart Association (NYHA) classification III or IV
* Severe coronary heart disease as manifest by a history of myocardial infarction or unstable angina in the last 6 months prior to visit 0
* Clinically significant cardiac valvular disease
* Subjects with an aortic aneurysm that, in the opinion of the investigator, will be unsuitable to be enrolled in the study.
* Type 1 diabetes mellitus (DM) or poorly controlled Type 2 DM as evidenced by glycosylated hemoglobin HbA1C of greater than 9% on visit 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-08 (Estimated); Study Completion 2019-12-08 (Estimated)

PRIMARY OUTCOMES:
Change in mean seated systolic blood pressure (MSSBP). | From baseline to treatment week 8

SECONDARY OUTCOMES:
Change in mean seated diastolic blood pressure (MSDBP). | From baseline to treatment week 8
Blood pressure Response Rate | Treatment week 8
  Response rate is defined as the percentage of subjects achieving a systolic blood pressure (SBP) response (MSSBP of < 140 mmHg or a reduction of MSSBP of > 20 mm Hg from baseline value), or a diastolic blood pressure (DBP) response (i.e. MSDBP of < 90 mmHg or a reduction of MSDBP of > 10 mm Hg from baseline value) after 8 weeks treatment.
Blood pressure Control Rate | Treatment week 8
  Control rate is the percentage of subjects that reach the predetermined blood pressure(BP) target < 140/90 mmHg. In addition, the percentage of subjects that reach the predetermined BP target < 140/90 mmHg for subjects without diabetes or chronic renal disorder(baseline estimated glomerular filtration rate(GFR) < 60 mL/min); <130/80 mmHg for subjects with diabetes or chronic renal disorder will be provided as well.
Mean change in systolic blood pressure and diastolic blood pressure in ambulatory blood pressure monitoring over 24 hours. | Treatment week 8
Number of participants with adverse events as a measure of safety and tolerability. | Treatment week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Italy (8):
  - Fondazione Università G.D'Annunzio, Chieti, Abruzzo
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - AAS 3 Friuli Alto Medio Collin, Udine, Friuli Venezia Giulia
  - Fondazione Salvatore Maugeri, Pavia, Lombardy
  - IRCCS Ist Neurologico Mediterraneo, Isernia, Molise
  - A.O.U. di Sassari, Sassari, Sardinia
  - A.O.U. Pisana, Pisa, Tuscany
  - AULSS 07 Pieve Soligo, Treviso, Veneto